CLINICAL TRIAL: NCT04383444
Title: Surveillance of Individuals Following SARS-CoV-2 Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200117; 20-I-0117
Record Dates: First submitted 2020-05-09; First posted 2020-05-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: COVID-19; Coronavirus; Antibody Testing; Severe Acute Respiratory Syndrome-Coronavirus-2 infection; Natural History
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 exposure: NIH staff exposed to SARS-CoV-2 or current or previous SARS-CoV-2 infection, but currently asymptomatic

SUMMARY:
Background:

People who have had contact with a person with a known SARS-CoV-2 infection are being told to self-quarantine for 14 days. This is done to avoid potential virus spread. But the actual time it takes for a person to develop an infection after being exposed to the virus is not well known. The proper quarantine time could be less or more than 2 weeks. Researchers hope this study can be used to help improve public health guidelines for quarantines, social distancing, and returning to work after a possible SARS-CoV-2 exposure.

Objective:

To better understand how long it takes a person to develop (or not develop) an infection with the SARS-CoV-2 virus after they have had contact with a person who has a confirmed infection.

Eligibility:

NIH staff members age 18 and older who had recent contact with a person who has a SARS-CoV-2 infection

Design:

Participants will have 3 study visits at the NIH Clinical Center. They may be asked to have an extra visit depending on the test results at the third visit.

At each visit, participants will give a blood and saliva sample. It will be used to test for SARS-CoV-2 antibodies. Their temperature will be taken. They will complete a short survey to collect data about possible COVID-19 symptoms. At the first visit only, they will also complete a survey that asks about their recent social contacts.

Two types of nasal samples will be collected at each visit. These samples will be tested for the SARS-CoV-2 virus.

1. a swab will be inserted deep into the back of the nose and
2. a swab will be inserted to the middle of your nose.

Participation lasts 3 to 4 weeks.

DETAILED DESCRIPTION:
Study Description:

This is a prospective longitudinal cohort study of individuals who have recently tested positive or are highly suspected to be positive for severe acute respiratory syndrome-coronavirus-2 (SARS-CoV- 2) infection. The aim is to correlate results of reverse transcription-polymerase chain reaction (RT-PCR) using various sample types, assays, and culture. We will enroll individuals with at least one recent positive RT-PCR test result (confirmed cases) and individuals whose referring physician highly suspects current or recent SARS-CoV-2 infection but the individual has not had access to testing (probable cases). At baseline, participants will undergo collection of nasopharyngeal (NP) swabs, saliva samples, and midturbinate swabs for SARS-CoV-2 RT-PCR and culture, and blood draw for antibody assay. Subjects enrolled as probable cases who have a positive baseline RT-PCR result and all subjects enrolled as confirmed cases (regardless of baseline result) will be followed with serial screenings until they have 2 consecutive negative RT-PCR test results.

Objectives:

Primary Objective:

Correlate results of SARS-CoV-2 RT-PCR using various sample types, antibody assays and culture.

Secondary Objectives:

1. Determine rate of culture positivity in individuals who persistently shed virus.
2. Correlate symptoms with culture positivity and RT-PCR cycle threshold.

Endpoints: Primary Endpoint: Results of SARS-CoV-2 RT-PCR using NP swab, saliva, and midturbinate swab, antibody assay and culture.

Secondary Endpoint:

1. SARS-CoV-2 culture and RT-PCR results.
2. Symptom checklist and RT-PCR cycle threshold value.

Study Population:

We will enroll up to 1,000 (accrual ceiling: 1,050) adults who have had one or more positive RT-PCR test result(s) within the last two weeks (confirmed cases) and those who have not been tested within the last two weeks but meet a high index of clinical suspicion for current or recent SARS-CoV-2 infection (probable cases).

Facilities Enrolling Participants:

NIH CC.

Study Duration: 3 years.

Participant Duration:

Probable cases who have negative RT-PCR results at baseline will have a single (baseline) visit. Probable cases with positive baseline RT-PCR and all confirmed cases will continue in the

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Able to attent study visits at the NIH.
2. Age greater than or equal to 18 years.
3. Meets one of the following case definitions:

   1. Confirmed case: At lease one current or recent (within past 14 days positive RT-PCR test for SARS-CoV-2.
   2. Probable case: Suspected current or recent (within the past 14 days) SARS-CoV-2 infection by referring physician but no availability of confirmatory test results.
4. Able to provide informed consent.
5. Willing to allow storage of samples for future research..

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. The most recent RT-PCR tests have yielded two negatives.
2. Inability or unwillingness to have NP sampling, mid-turbinate, or saliva sampling
3. Inability or unwillingness to have blood sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NIH staff or contractors working at an NIH facility and able to come to the NIH campus for study visits.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Results of SARS-CoV-2 RT- PCR testing, antibody assay, and culture | Days 1, 14, then every 2-4 weeks as needed
  Correlate results of SARS-CoV-2 RT-PCR using various sample types, antibody assays, and culture.

SECONDARY OUTCOMES:
SARS-CoV-2 culture and RT-PCR results | Days 1, 14, then ever 2-4 weeks as needed
  Determine rate of culture positivity in individuals who persistently shed virus.
Symptom checklist and RT-PCR cycle threshold | Days 1, 14, then every 2-4 weeks as applicable
  Correlate symptoms with culture positivity and RT-PCR cycle threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Holland, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0117.html

DOCUMENTS (1):
  • Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT04383444/ICF_000.pdf